CLINICAL TRIAL: NCT07356076
Title: The Use of Electrical Impedance Tomography (EIT) in Pulmonary Diseases
Status: Recruiting | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Collaborators: Brno University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: OP JAK ITI VZ 3; CZ.02.01.01/00/23_021/0008829 (Other Grant/Funding Number: Operational Programme Jan Ámos Komenský financed by the European Union (EU) and the State Budget of Czech Republic)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lung Diseases
Keywords: Electrical Impedance Tomography; Spirometry; Lung Diseases; Lung Assessment
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with lung diseases: Adults aged 18 years and older
  Individuals diagnosed with any of the following lung diseases, as these are the primary focus of the study: Chronic obstructive pulmonary disease, Asthma, Pulmonary fibrosis, Pneumonia, Patients with a history of COVID-19 infection showing residual pulmonary findings.
  Ability to perform spirometry while seated, except for possible participants who are specifically part of a subgroup analysis where inability to perform spirometry is the condition which is studied.
  Signing of an informed consent that has been approved by the ethics committee
- Healthy controls: Adults aged 18 years and older
  Healthy subjects will be enrolled to obtain normal standard values (with normal physical examination and no respiratory symptoms, BMI 18-31 - cause EIT performance can be BMI dependent, Non-smokers or ex-smokers abstinent ≥12 months)
  Ability to perform spirometry while seated, except for possible participants who are specifically part of a subgroup analysis where inability to perform spirometry is the condition which is studied.
  Signing of an informed consent that has been approved by the ethics committee

SUMMARY:
The study titled "The Use of Electrical Impedance Tomography (EIT) in Pulmonary Diseases" investigates the impact of using EIT as a non-invasive method to monitor the distribution of pulmonary ventilation and its relationship to standard spirometry in patients with various lung diseases. The main aim of this study is to investigate new approaches to the assessment of lung status and diagnosis of lung diseases.

Unlike spirometry, which has long been a well-known and important diagnostic tool in pulmonary medicine, and which provides valuable information about the volume and flow of inspired and expired air, EIT provides spatial information about the distribution of ventilation in real time and without the need for active patient cooperation. Research and practice have shown that spirometry is problematic in specific groups of patients, such as patients with tracheostomy or facial palsy. The technology should also enable detection of the disease in its early stages, when treatment is most effective.

300 participants in the experimental group and 100 participants in the control group will receive spirometry and electrical impedance tomography independent examination.

The primary endpoint of the study is to investigate the potential of EIT in respiratory medicine, specifically identifying the relationship between EIT and traditional spirometry. This effort is motivated by the need for novel noninvasive methods for the diagnosis and monitoring of respiratory diseases, especially in patients unable to undergo conventional spirometry, or in case of interventions requiring real-time feedback. The purpose of the research project in relation to these objectives is to bring new possibilities in the field of diagnosis and monitoring of lung diseases through EIT, which could lead to significant improvements in patient care.

Demographic and anthropometric data, including age, sex, body height, body weight, body mass index (BMI), chest circumference, and smoking history will be collected in all participants. These parameters will be used as covariates in the analysis to assess their impact on EIT-derived indicators and to improve normalization of EIT signals.

Additionally, the study aims to develop and validate a machine learning model, particularly a deep neural network, capable of predicting standard spirometric parameters (e.g., FEV1, FVC, PEF) based solely on EIT signals. This could allow for an accurate assessment of dynamic pulmonary volumes in cooperating patients who are unable to undergo conventional spirometry (e.g. patients with tracheostomy).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Individuals diagnosed with any of the following lung diseases, as these are the primary focus of the study: Chronic obstructive pulmonary disease, Asthma, Pulmonary fibrosis, Pneumonia, Patients with a history of COVID-19 infection showing residual pulmonary findings.
* Additionally, healthy subjects will be enrolled to obtain normal standard values (with normal physical examination and no respiratory symptoms, BMI 18-36 - cause EIT performance can be BMI dependent, Non-smokers or ex-smokers abstinent ≥12 months)
* Ability to perform spirometry while seated, except for possible participants who are specifically part of a subgroup analysis where inability to perform spirometry is the condition which is studied.

Signing of an informed consent that has been approved by the ethics committee

Exclusion Criteria:

* Patients under 18 years of age
* Severe cardiovascular disease
* Pregnancy
* Inability to express consent
* Acute respiratory infection: Except for those recovering from pneumonia or COVID-19 within the study focus, participants with current respiratory infections will be excluded to avoid confounding effects on lung function tests
* Inability to perform spirometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the Department of Pulmonary Diseases and Tuberculosis, University hospital Olomouc, and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between EIT-derived FEV1 and spirometry-derived FEV1 | At baseline visit (single measurement)
  Comparison of forced expiratory volume in 1 second predicted from EIT using a trained neural network with direct spirometry measurement.
  Metric: Mean Absolute Error (MAE), Bland-Altman limits of agreement, Pearson correlation coefficient (r)

SECONDARY OUTCOMES:
Forced Expiratory Volume in One Second (FEV1) | At baseline visit (single measurement)
  FEV1 represents the volume of air that can be forcibly exhaled in the first second of a forced exhalation Measurements will be performed using calibrated spirometry. FEV1 is a standard measure of pulmonary function.
  Unit of Measure: Liters
Forced vital capacity (FVC) | At baseline visit (single measurement)
  FVC represents the largest amount of air that can be forcefully exhaled from maximum inspiration.
  Unit of Measure: Liters
Peak Expiratory Flow (PEF) | At baseline visit (single measurement)
  PEF represents the maximum flow achieved during forceful exhalation from maximum inspiration and is a reliable indicator of ventilation adequacy as well as airflow obstruction.
  Unit of Measure: Liters/minute
Estimated Lung Age (ELA) | At baseline visit (single measurement)
  ELA is a calculation that estimates the age of a person's lungs based on their lung function, particurarly FEV1 (forced expiratory volume in one second), compared to normal lung function for their chronological age. Secondary objectives include comparison of regional ventilation patterns from EIT with spirometric flow-volume loop abnormalities, assessment of EIT-based estimated lung age, and determination of EIT's ability to track treatment response over time.
Forced Expiratory Volume in Three Seconds (FEV3) | At baseline visit (single measurement)
  FEV3 represents the volume of air that can be exhaled during the first three seconds of forceful exhalation after maximum inspiration.
  Unit of Measure: Liters
Forced Expiratory Volume in Six Seconds (FEV6) | At baseline visit (single measurement
  FEV6 represents the volume of air that can be exhaled during the first six seconds of forceful exhalation after maximum inspiration
  Unit of Measure: Liters
FEV1/FVC ratio | At baseline visit (single measurement
  FEV1/FVC is the ratio of forced expiratory volume in one second to forced vital capacity.
  Unit of Measure: Percentage
Forced Expiratory Flow at 50 % of FVC (FEF50) | At baseline visit (single measurement
  FEF50 is the flow rate at the 50% point of the total volume (FVC) exhaled.
  Unit of Measure: Liters
Forced Expiratory Flow at 75 % of FVC (FEF75) | At baseline visit (single measurement
  FEF75 is the flow rate at the 75% point of the total volume exhaled.
  Unit of Measure: Liters

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary Diseases and Tuberculosis, University hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Undecided